CLINICAL TRIAL: NCT03905187
Title: A Perspective Randomized Study of Impact of Stress Management Involved Cardiac Rehabilitation on Psychological States and Clinical Outcomes of Patients After Acute Myocardial Infarction or Heart Failure
Brief Title: Stress Management Modified Cardiac Rehabilitation in Patients After Acute Myocardial Infarction or Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jing Ma (Other)
Responsible Party: Sponsor-Investigator, Jing Ma, Clincial professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 301CRS20181228
Record Dates: First submitted 2019-02-03; First posted 2019-04-05 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Acute Myocardial Infarction; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): Group received education only
  Interventions: Behavioral: Education
- Traditional CR Group (Other): Group received cardiac rehabilitation including education and exercise
  Interventions: Behavioral: Traditional CR
- Stress-Modified CR Group (Experimental): Group received cardiac rehabilitation including education, exercise and stress management
  Interventions: Behavioral: Modified CR

INTERVENTIONS:
Behavioral: Modified CR — Stress management involved modified cardiac rehabilitation
  Arms: Stress-Modified CR Group
Behavioral: Traditional CR — Traditional cardiac rehabilitation
  Arms: Traditional CR Group
Behavioral: Education — Education
  Arms: Control Group

SUMMARY:
The purposes of this study is to evaluate the improvement of a stress management involved cardiac rehabilitation program on the psychological states, quality of life and clinical outcomes of patients after acute myocardial infarction or heart failure.

DETAILED DESCRIPTION:
The purposes of this study is to evaluate the improvement of a stress management involved cardiac rehabilitation program on the psychological states, quality of life and clinical outcomes of patients after acute myocardial infarction or heart failure. The investigators performed modified cardiac rehabilitation program involving stress management on the patients who suffered from acute myocardial infarction or severe heart failure who were admitted to the CCU. Then the psychological states, quality of life and clinical outcomes were followed up.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old with a diagnosis of AMI (include ST segment elevated myocardial infarction and non-ST segment elevated myocardial infarction) or heart failure

Exclusion Criteria:

* Uncontrolled tachycardia (heart rate at rest >120bpm
* Uncontrolled polypnea（breath rate at rest >30 breath per minute
* Uncontrolled respiratory failure （SPO2 ≤90%）
* Uncontrolled hypertension （pre-exercise SBP>180mmHg or DBP>110mmHg）
* Weight change in 72 hours >1.8kg
* Uncontrolled hyperglycemia (Random blood glucose>18mmol/L)
* Uncontrolled malignant arrhythmia with hemodynamic instability
* Unoperated pseudoaneurysm、artery dissection
* Uncontrolled septic shock and septicopyemia
* Unoperated severe valvular heart disease or acute phase of heart failure caused by myocardial heart disease
* nervous system disease, motor system diseases and rheumatic diseases considered possibly worsened by exercise
* Uncooperation of the patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-04-16 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
The score of anxiety test questionnaire decreased | 6 month
  The score of anxiety test questionnaire(Generalized Anxiety Disorder,GAD-7, normal range 0-21, partially reflecting the severity of anxiety with the higher score) decreased
The score of Medical Outcomes Study Questionnaire Short Form 36 Health Survey (36-Item Short Form Survey) increased | 6 month
  The score of Medical Outcomes Study Questionnaire Short Form 36 Health Survey (abbreviation form is 36-Item Short Form Survey) increased. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability, The sections consists of Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, and Mental health. The total score of SF 36 Health survey is higher, the quality of life is higher.
The score of patient health questionnaire decreased | 6 month
  The score of patient health questionnaire (PHQ9, normal range 0-27，indicating the profile of depression with the higher score) decreased
The score of Chinese perceived stress scale decreased. | 6 month
  The score of Chinese perceived stress scale (CPSS, 0-56, higher means more stress) decreased.

SECONDARY OUTCOMES:
incidence of MACE in patients after acute myocardial infarction | 6 month
  any incidence of the following: death, cardiac death, AMI, revascularization, stroke
incidence of MACE in patients with heart failure | 6 month
  death, cardiac death, resynchronization
improvement of exercise capacity | 6 month
  6 minute walking distance
incidence of rehospitalization | 6 month
  incidence of rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, Principal Investigator — Department of Cardiology in Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: The IPD of the publication will be shared, including characteristic data, results, clinical follow up data.